CLINICAL TRIAL: NCT07137676
Title: Monitoring and Cognitive Appraisal: The Etiology of Psychological Disorders and The Divergence Between Behavioural and Self-reported Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Principal Investigator, Leon Alker, Chief Clinical Neuropsychologist (Winterberg, Germany), St. Franziskus Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: file reference 2024-01k; ethics comittee (Other: St. Franzikus Hospital Winterberg)
Record Dates: First submitted 2025-07-25; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Geriatric Patients in a Pre-rehabilitative Treatment; Mild Cognitive Impairment (MCI)
Keywords: monitoring; cognitive appraisal
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AX-CPT Treatment (Experimental): Treatment with the AX-CPT
  Interventions: Behavioral: AX-CPT
- Control Group (Other): AX-CPT is merely administrated as pre-and posttest measure.
  Interventions: Other: No Interventions

INTERVENTIONS:
Behavioral: AX-CPT — administration of the AX-CPT
  Arms: AX-CPT Treatment
Other: No Interventions — Control group with no intervention treatment
  Arms: Control Group

SUMMARY:
The study investigates the etiology of psychogical disorders from a neuropsychological perspective based on monitoring and cognitive appraisal.

ELIGIBILITY:
Inclusion Criteria:

* geriatric patient of the St. Franziskus-Hospital, Germany.

Exclusion Criteria:

* severe dementia
* delirium
* psychotic disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-16 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
AX-CPT (AX-Continuous Performance Test) | from beginning (day 2) of the hospitalization to the end (day 14) of the biweekly pre-rehabilitative treatment.
  The AX-CPT assesses cognitive control through error rates and reaction times. Range: Error rate: 0-100%; Reaction time: measured in milliseconds Interpretation: Lower error rates and faster reaction times indicate better cognitive control performance.
CCFQ (Cognitive Control and Flexibility Questionnaire) | Day 1 (pretest) and Day 14 (posttest)
  The CCFQ measures self-reported cognitive flexibility and control.
  Scale title: Cognitive Control and Flexibility Questionnaire Range: 1-7 per item Interpretation: Higher scores indicate greater cognitive flexibility and control.
BSI-18 (Brief Symptom Inventory - 18) | Day 1 (pretest) and Day 14 (posttest)
  T he BSI-18 assesses psychological symptom severity in terms of depression, anxiety, and somatization.T
  Scale title: Brief Symptom Inventory - 18 Range: 0-4 per item Interpretation: Higher scores indicate greater symptom severity.
MHC-SF (Mental Health Continuum - Short Form) | Day 1 (pretest) and Day 14 (posttest)
  Measures emotional, psychological, and social well-being. Range: 1-6 per item Interpretation: Higher scores indicate better mental health.

SECONDARY OUTCOMES:
General Self-Efficacy assessed via General Self-Efficacy Scale (SWE) | Day 1 (pretest) and Day 14 (posttest)
  Evaluation of perceived self-efficacy across various life domains. Range: 1-4 per item Interpretation: Higher scores indicate greater self-efficacy.
Treatment Beliefs assessed via Palermo Questionnaire | Day 1 (pretest) and Day 14 (posttest)
  Beliefs and expectations regarding treatment effectiveness. Range: 1-5 per item Interpretation: Higher scores indicate stronger and more positive treatment beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Franziskus-Hospital Winterberg, Winterberg, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
the data contains patient-relevant information that is protected under the European General Data Protection Regulation act.